CLINICAL TRIAL: NCT06027697
Title: Prospective Evaluation of Subchondroplasty in Advanced Knee Osteoarthritis.
Status: Not yet recruiting | Type: Observational
Sponsor: Clinique Paris-Bercy (Other)
Collaborators: CEISO (Industry); ClinServ (Unknown)
Responsible Party: Sponsor
Other Study IDs: Subchondroplasty
Record Dates: First submitted 2023-08-31; First posted 2023-09-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-08

CONDITIONS: Knee Osteoarthritis
Keywords: Knee osteoarthritis; Subchondroplasty; Knee mechanical pain; AccuFill Porous Bone Substitute Material; Minimally invasive surgical procedure
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subchondroplasty: AccuFill Porous Bone Substitute Material (BSM) will be administrated to the patient during a subchondroplasty procedure (treatment visit).
  During the inclusion visit and the follow-up visits (Week 3, Week 6; Month 3, Month 6, Month 12, Month 24, Month 36, Month 48) the doctor will proceed the usual clinical exam and the patients will fulfil the validated questionnaires and scales to assess pain, functional impairments and subjective improvement.
  Interventions: Device: AccuFill® Porous Bone Substitute Material (BSM)

INTERVENTIONS:
Device: AccuFill® Porous Bone Substitute Material (BSM) — The patient will undergo a minimally invasive surgery procedure (subchondroplasty) to receive the medical device AccuFill® Porous Bone Substitute Material (BSM).
  Other Names: Subchondroplasty

SUMMARY:
The goal of this observational study is to evaluate the technique of subchondroplasty in patients with advanced knee osteoarthritis.

The main question it aims to answer is:

• Does the subchondroplasty technique with the administration of AccuFill Porous Bone Substitute Material (BSM) is effective in the relief of mechanical pain in patient with knee osteoarthritis ?

Participants will go under a minimally invasive surgery procedure (subchondroplasty) and fulfil 3 validated questionnaires to assess pain, functional impairments and subjective improvement.

This study will be conducted for 4 years.

DETAILED DESCRIPTION:
Background :

The technique of subchondroplasty is recent and was created to follow the availability of low-viscosity injectable phosphocalcic cement. It is aimed at osteoarthritic lesions and proposes to treat subchondral disease associated with the process of osteoarthritic degeneration, and which would be particularly painful in the support area.

This technique seems interesting in terms of effectiveness with less risk since it is a minimally invasive percutaneous procedure and it is systematically practiced on an outpatient basis.

In this context, the principal investigator has decided to conduct a long-term study for the first time in France in order to collect clinical data and data on the safety profile of the device.

Design :

This study is prospective, longitudinal, observational, single-arm, open monocentric and is a post-market study.

Intervention :

As the current study is observational, the study will follow the usual standard of care.

The participation of the patient can be divided in 2 parts :

* The first part is the treatment. After the inclusion of the patient, this latest will undergo a minimally invasive surgery procedure (subchondroplasty) to receive the treatment (AccuFill Porous Bone Substitute Material (BSM)).
* The second part is the follow-up visits. During this part the patient will follow a appointment schedule with the doctor in order for the physicien to realised a clinical examination and for the patient to fulfil the 3 validated questionnaires. These visits will be spaced out over 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years of age or older;
* Patient with a Body Mass Index ≤35 (BMI=kg/m2);
* Patient with Kellgren-Lawrence grade 3-4 Osteoarthritis, as reviewed on MRI and plain radiography;
* Patient with knee bone marrow lesions confirmed by MRI result at least 3 months before the intervention;
* Patients with degenerative knee pathology at the prosthetic stage (outdated medical treatments), with a frontal deformity of less than 12°, (and wishing to avoid or delay the prosthetic procedure as much as possible) / goniometry);
* Patient with unbearable mechanical pain with a walking perimeter limited at 500 m
* Patient with non-surgical treatment failure (infiltration of Platelet Rich Plasma (PRP), corticoids, acid hyaluronic);
* Patient who agrees to participate in the study and who signed the informed non-opposition form;
* Patient physically and mentally willing and able, in the Investigator's opinion at the time of enrolment, to be compliant with the protocol including all follow-up visits, survey completion, weight- bearing restrictions, and post-operative rehabilitation;
* Patient with social protection.

Exclusion Criteria:

* Patient with a Body Mass Index > 35 (BMI=kg/m2);
* Patient with inflammatory rheumatic pathologies;
* Patient with frontal deformities (varus, valgus) of more than 12°;
* Patient with degenerative pathologies at the operative stage but likely to benefit from a conservative intervention (osteotomy), except if the knee is centred;
* Patient with stiff knees (more than 20° of flexum and/or less than 90° of flexion);
* Patient with painful severe femoro-patellar osteoarthritis;
* Patient with contraindications for Magnetic Resonance Imaging (MRI);
* Patient with history of systemic diseases which could contribute to secondary arthropathies (e.g., sickle cell disease, hemochromatosis, or autoimmune disease);
* Patient with history of cognitive-behavioural disorders that could interact with assessment by self-questionnaire;
* Patient with local or general infection or suspicion of infection;
* Patient with severe coagulation disorders;
* Patient with primary bone tumour in the knee area,
* Patient with undercurrent serious pathology with life expectance < 2 years;
* Female patient of childbearing age that are known to be pregnant during inclusion visit or wishing to become pregnant before treatment;
* Patient who has forfeited their freedom by administrative or legal award, or is under guardianship or under limited judicial protection;
* Patient participating in another interventional clinical trial or testing an experimental drug within 30 days of inclusion in the study;
* Patients who cannot read or write French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who go for a consultation for refractory mechanical knees pain
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline (inclusion) in Patient-Reported Pain Scores on the Visual Analog Scale (VAS) to 3 months. | Month 3
  Visual Analog Scale (VAS) is a unidimensional measure of pain intensity, used to record patients' pain progression. It will helped the patient to assess the perceived mechanical knee pain on a horizontal, non-calibrated line of 10 cm, ranging from very low (0) to very high (10)

SECONDARY OUTCOMES:
Change from baseline (inclusion) in Patient-Reported Pain Scores on the Visual Analog Scale (VAS) to each visits | Week 3, Week 6, Month 6, Month 12, Month 24, Month 36, Month 48
  Visual Analog Scale (VAS) is a unidimensional measure of pain intensity, used to record patients' pain progression. It will helped the patient to assess the perceived mechanical knee pain on a horizontal, non-calibrated line of 10 cm, ranging from very low (0) to very high (10).
Change from baseline (inclusion) in International Knee Documentation Committee (IKDC) score to each visits | Week 3, Week 6, Month 3, Month 6, Month 12, Month 24, Month 36, Month 48
  IKDC is a subjective knee evaluation form to detect improvement or deterioration in symptoms, function and sports activities due to knee impairment.
  This self-questionnaire is divided into three parts (symptoms, sports activities, function) and gives a score between 0 (worst) and 100 (best).
Change from baseline (inclusion) for the Knee injury and Osteoarthritis Outcome Score (KOOS) to each visits | Week 3, Week 6, Month 3, Month 6, Month 12, Month 24, Month 36, Month 48
  KOOS is a knee-specific instrument, developed to assess the patient's opinion about their knee and associated problems. The KOOS evaluates both short-term and long-term consequences of knee injury.
  It contains 42 items divided into five subscales:
  KOOS Pain, KOOS Symptoms, Activities of Daily Living (KOOS ADL), Sport (KOOS Sport), and Quality of Life regarding the knee (KOOS QOL). Total scores can range from 0 to 100.
Rate of adverse events | Week 3, Week 6, Month 3, Month 6, Month 12, Month 24, Month 36, Month 48
  To assess the rate of adverse events
Radiography and MRI evolution of the knee lesions from baseline (inclusion) to 24 months | Month 24
  Morphologic evolution of knee joint on MRI and radiography
Rate of conversion to prosthetic replacement | Month 12, Month 24, Month 36, Month 48
  Rate of patient who have to undergo to prosthetic replacement

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Paris Bercy, Charenton-le-Pont, France